CLINICAL TRIAL: NCT06425042
Title: Boosting the NAD+ Levels in Older Individuals Via Nicotinamide Riboside Supplementation and Exercise Training to Promote Metabolic Health
Brief Title: Nicotinamide Riboside Supplementation and Exercise Training to Promote Healthy Longevity
Acronym: RESTORENAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Finis Terrae University (Other)
Responsible Party: Principal Investigator, Rodrigo Mancilla, Doctor, PhD, Finis Terrae University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-041
Record Dates: First submitted 2024-05-14; First posted 2024-05-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Healthy Aging; Lifestyle-related Condition; Metabolic Diseases
MeSH Terms: conditions — Mental Disorders; Metabolic Diseases | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NR+EXTR (Experimental): This arm will ingest NR orally and perform exercise training
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- PLA+EXTR (Placebo Comparator): This arm will ingest placebo orally and perform exercise training
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — Participants will ingest 1g/d of NR orally during 12 weeks in parallel to a exercise training program
  Arms: NR+EXTR
Dietary Supplement: Placebo — Participants will ingest 1g/d of placebo orally during 12 weeks in parallel to a exercise training program
  Arms: PLA+EXTR

SUMMARY:
The prevalence of age-related chronic diseases (like obesity, type 2 diabetes and cardiovascular diseases) is mounting worldwide, reaching pandemic proportions. These age-related chronic diseases are associated with diminished skeletal muscle mitochondrial function in humans. Nicotinamide adenosine dinucleotide (NAD) is a coenzyme that regulates mitochondrial function, therefore, plays an important role in energy metabolism. Importantly, it has been shown that high cellular NAD+ levels as well as a high NAD+/NADH ratio promote metabolic and mitochondrial health. In contrast, NAD+ bioavailability declines upon aging in humans as well as in animal models of metabolic disorders and type 2 diabetes. These findings fuel the notion of boosting the NAD+ bioavailability in order to improve metabolic disturbances and mitochondrial dysfunction in aged individuals. Supplementation with nicotinamide riboside (NR), a naturally occurring form of vitamin B3, boosts cellular NAD+ levels. However, in contrast to animal studies, NR supplementation in humans has so far been unsuccessful in improving skeletal muscle mitochondrial function, exercise capacity or insulin sensitivity. Interestingly, Recently, it has been suggested that metabolic conditions where NAD+ levels become limited, is needed for NR supplementation to exert beneficial health effects. This metabolic condition could be achieved by exercise. However, studies combining NR and exercise are lacking, and that is why we will perform the present study.

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to provide signed and dated written informed consent prior to any study specific procedures
* Aged ≥ 60 and ≤ 80 years
* Body mass index (BMI) 25 - 35 kg/m2
* Stable dietary habits (no weight loss or gain > 5 kg in the past 3 months)
* No signs of active cardiovascular disease, liver or kidney malfunction

Exclusion Criteria:

* Patients with congestive heart failure and and/or severe renal and or liver insufficiency
* Uncontrolled hypertension
* Any contra-indication for MRI scanning
* Alcohol consumption of > 3 servings per day for man and >2 servings per day for woman
* Smoking
* Unstable body weight (weight gain or loss > 5kg in the last 3 months)
* Engagement in structured exercise activities > 2 hours a week
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the Investigator which would possibly hamper our study results
* Use of food supplements containing NR or Resveratrol (similar working mechanisms)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle mitochondrial respiratory capacity | 12 weeks
  Skeletal muscle mitochondrial respiratory capacity will be measured in permeabilized fibres.

SECONDARY OUTCOMES:
Quantification of proteins that regulate oxidative metabolism | 12 weeks
  Quantification of proteins content of oxidative phosphorylation system in muscle biopsies
Skeletal muscle mitochondrial content | 12 weeks
  Proteins content of oxidative phosphorylation system will be quantified from muscle biopsy
Maximal aerobic capacity | 12 weeks
  Maximal aerobic capacity will be measure upon a progressive cycling test
Walking speed and distance | 12 weeks
  Walking speed and distance will be measured via the 6-minutes walking test
Seating and standing transitions | 12 weeks
  Time spent on performing seating and standing transitions will be measured upon the timed-up and go test
Exercise efficiency | 12 weeks
  Exercise efficiency will be measured upon a sub maximal cycling test and indirect calorimetry
Intrahepatic liver fat content | 12 weeks
  Intrahepatic liver fat content will be measured by 1H-MRS
Body weight | 12 weeks
  body weight will be measured in kilograms
Total muscle mass | 12 weeks
  total muscle mass will be measured in kilograms and/or percentage
Total fat mass | 12 weeks
  Total fat mass will be measured in kilograms and/or percentage
Fat-free mass | 12 weeks
  Fat-free mass will be measured in kilograms and/or percentage
NAD+ levels | 12 weeks
  NAD+ levels in circulation and in skeletal muscle
24h Blood pressure | 12 weeks
  24h Blood pressure will be measured with a continuous blood pressure holder device
Resting energy expenditure | 12 weeks
  Resting energy expenditure will be measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Finis Terrae University, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No